CLINICAL TRIAL: NCT03740815
Title: Assessment of the Feasibility of Ultrasound Guided Serratus Plane Block Associated With Sedation as Anesthetic Technique in Axillary Dissection
Brief Title: Feasibility of Serratus Plane Block Associated With Sedation in Axillary Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 89037818.0.0000.5274
Record Dates: First submitted 2018-06-25; First posted 2018-11-14 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia; Regional Anesthesia Morbidity; Axillary Metastases; Nerve Block; Analgesia; Skin Cancer
MeSH Terms: conditions — Agnosia; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serratus plane block plus sedation (Experimental): Serratus plane block plus intravenous sedation as anesthetic technique during axillary dissection procedure.
  Interventions: Procedure: Serratus plane block; Procedure: Axillary dissection; Procedure: Intravenous sedation

INTERVENTIONS:
Procedure: Serratus plane block — Ultrasound guided injection of local anesthetic between latissimus dorsi and serratus muscles at mid axillary line.
Procedure: Axillary dissection — Axillary dissection is a surgical procedure that incises the axilla to identify, examine, or remove lymph nodes.
  Other Names: Axillary limphadenectomy
Procedure: Intravenous sedation — Administration of sedatives thru an intravenous access to achieve relaxion and improve operative conditions.
  Other Names: Sedation

SUMMARY:
INTRODUCTION: The axillary lymphadenectomy procedure is known to be associated with late postoperative complications, such as chronic pain and changes in shoulder mobility. Recently, several thoracic ultrasound guided interfascial blocks have been described, including serratus plane block. These blocks were associated with reduced postoperative pain scores in breast surgeries but were never evaluated in axillary dissection. The safety and feasibility of performing axillary dissection under local anesthesia and tumescent anesthesia associated with sedation has been demonstrated in case series, although it is not already the standard technique.

DISCUSSION: This project aims to investigate the feasibility of the serratus plane block associated with intra-venous sedation in a prospective case series including 15 patients submitted to axillary dissection, by scoring patient and surgeon satisfaction with the technique, pain, quality of life with EORTC QLQ-C30 questionnaire, and quality of recovery with QoR-40 questionnaire in the first 30 postoperative days.

DETAILED DESCRIPTION:
This study is a prospective case series. All patients should go through a preoperative evaluation with an anesthesiologist. At that time the eligibility for the study will be evaluated and if the patient consent to participate in the study.

The following parameters shall be evaluated in the ambulatory evaluation:

* Age
* Anthropometric data (weight and height);
* Presence of comorbidities;
* Revised cardiac index (LEE);
* Estimation of functional capacity in metabolic equivalents (METs) by history;
* Performance Status by the scale of Eastern Cooperative Oncology Group (ECOG);
* Determination of the physical status by the American Society of Anesthesiologists (ASA) classification;
* QoR-40 recovery quality scale, validated for Brazilian Portuguese;
* Quality of life EORTC QLQ-C30 questionnaire, validated for Brazilian Portuguese.

During the anesthetic procedure, the following standard technique should be applied: peripheral venous access, dipyrone 30 mg/kg, antibiotic according to the institutional protocol, moderate sedation with intravenous propofol in continuous infusion in the absence of any contraindication. Midazolam will be used in case of contraindication to propofol or during the execution of the block according to preference of the researcher who will perform the block. Associated with propofol infusion, the alpha agonist dexmedetomidine may be used in continuous infusion associated with fentanyl, tramadol, dextroketamine, magnesium sulfate, dipyrone and tenoxicam, whose uses will be evaluated on a case-by-case basis and will be recorded in the database.

In case of conversion to general anesthesia, the airway control should be carried out preferably with laryngeal mask, with the orotracheal intubation as an alternative option. The maintenance of anesthesia will be in this case using propofol continuous infusion in the absence of contraindications, otherwise sevoflurane will be used. Postoperative nausea and vomiting prophylaxis will be done with four milligrams of dexamethasone and ondansetron.

Patients will be submitted serratus plane block according to the technique described in Blanco. The patients will be positioned in a supine position. The transducer of the ultrasound device is protected with sterile cover. The ultrasound probe is positioned in the mid clavicular region of the thoracic wall in a sagittal plane. Using a nether-lateral path with the probe, will be counted the ribs, until the fifth rib is identified in the mid axillary line. In this position, over the fifth rib, the latissimus dorsi muscle superficially and the serratus muscle deeper and lower can be easily observed. The identification of the thoracodorsal artery with use of doppler imaging assists in identifying the superficial plane to the serratus muscle. Once identified the structures, the needle is introduced in the plane of the transducer positioning its tip on the surface of the serratus muscle. Then 40 ml of solution with 1% lidocaine, adrenaline 1:200,000 and ropivacaine 0.5% are injected in patients above 50kg and 32ml of the same solution in patients with body weight between 40 and 50kg aiming to respect the maximum dose of local anesthetic recommended.

At the end of the surgical procedure the patient will be referred to the anesthetic recovery unit. The extension of the blockade will be then evaluated. They will be discharged to ward as soon as they get the discharge criteria.

The surgical time, time for execution of the blockage (counted from the placement of the sterile field until the removal of the needle), the surgical room time, estimated bleeding, presence of surgical complications or anesthetic and number of lymph nodes extracted will be registered. At the end of the surgery the surgeon will be asked to fill out a range of Likert 5 points on his opinion on the quality of anesthesia (extremely satisfied, satisfied, not satisfied or dissatisfied, dissatisfied, extremely dissatisfied) and to compare the quality of anesthesia with general anesthesia on a 3-point scale (indistinguishable from general anesthesia, sufficient to perform the procedure, extremely challenging/inadequate).

On the first day of postoperative the standard analgesia will be carried out with dipyrone 30 mg/kg IV every 4 hours, associated with tenoxicam 20mg every 12 hours. In case of contraindication to dipyrone, will be administered paracetamol 500 mg VO every 6 hours. As a rescue therapy the default option is tramadol 50mg IV up to every 4 hours (daily maximum dose of 300mg/day and morphine 4 mg each hour (in case of allergy or intolerance to tramadol and rescue the tramadol). If necessary more than 24 hours of hospitalization, postoperative analgesia will be performed as option of the assistant team. The use of postoperative painkillers will be recorded in the database.

All patients should be evaluated on the first postoperative day with record of the verbal numerical scale for the evaluation of pain at rest, cough and abduction of 90 Degrees of the member and the presence of adverse effects. They be asked to fill the scale of Likert of 5 points with his opinion on the quality of anesthesia (extremely satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, extremely dissatisfied) and the scale of recovery quality QoR-40. Between the twenty-eighth and the thirtieth-fifth postoperative day All patients will be reassessed, occasion where the scale of recovery quality QoR-40 and the scale of quality of life EORTC QLQ-C30, presence of surgical wound infection will be applied, cutaneous necrosis, seroma, lymphedema, lymphatic fistula and date of drain removal.

ELIGIBILITY:
Inclusion Criteria:

* Undergo axillary dissection due to metastatic skin or soft tissue cancer;
* ASA physical status classification between I and III;
* have signed the informed consent.

Exclusion Criteria:

* weight less than 40 kilograms;
* tumor affecting topography to be blocked;
* presence of ulcerated lesion in the axilla;
* presence of coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who needed conversion to general anesthesia | Intraoperative
  Percentage of patients who needed conversion to general anesthesia. A percentage from 0 to 100%, where 0% means that no patient needs technique conversion to general anesthesia and 100% means that all patients need it.

SECONDARY OUTCOMES:
The 30-item European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire. | Preoperative and in Postoperative day 30
  The QLQ-C30 is composed of multi-item scales and single-item measures. These include:
  * A global health status / QoL scale
  * Five functional scales (Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning)
  * Three symptom scales (Fatigue, Nausea and vomiting, Pain)
  * Six single items (Dyspnoea, Insomnia, Appetite loss, Constipation, Diarrhoea, Financial difficulties) Each of the multi-item scales includes a different set of items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems . The scales are scored as described as described in EORTC QLQ-C30 Scoring Manual. 2001 EORTC, Brussels.
QoR-40 questionnaire | Preoperative, First postoperative day visit and in Postoperative day 30
  Quality of Recovery - 40 Item questionnaire
  QoR-40 score is a score developed to estimate the quality of recovery after anesthesia. It consists of a 40-item questionnaire with items on a five- point Likert scale (for positive items, 1 'none of the time' to 5 'all of the time'; for negative items the scoring was reversed). It is scored as follows:
  QoR-40 dimensions
  * Emotional state (9-45)
  * Physical comfort (12-60)
  * Psychological support (7-35)
  * Physical independence (5-25)
  * Pain (7-35) Global QoR-40 (40-200)
Surgeon satisfaction - 5 points Likert scale | Imediate postoperative period
  A five points Likert scale will be applied to the main surgeon responsible for the operation.
  The surgeon will be asked to fill out a Likert 5 points scale to access his opinion about the quality of anesthesia (extremely satisfied, satisfied, not satisfied or dissatisfied, dissatisfied, extremely dissatisfied).
Patient satisfaction - 5 points Likert scale | First postoperative day visit
  A five points Likert scale will be applied to the patient in the first postoperative day visit to access his opinion about the quality of the anesthesia (extremely satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, extremely dissatisfied).
Numeric pain rating scale (0-10) | Preoperative, postoperative day 1 and 30
  Eleven point numeric pain rating scale (0 means no pain and 10 means worst possible pain).
Analgesic requirement | Intraoperative and postoperative day one (cumulative dose)
  All the anesthetics and analgesics used in intraoperative and postoperative period will be recorded. Doses will be recorded in database.
Number of lymph nodes extracted | Postoperative day 30 (according to anatomopathological report)
  Number of lymph nodes extracted according to anatomopathological report.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Theobald, MD, Principal Investigator — National Cancer Institute of Brazil (INCA - Brazil)
Locations (1):
- Hospital do Câncer II - National Cancer Institute of Brazil (INCA - Brazil), Rio de Janeiro, Rio de Janeiro/RJ, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fecho K, Miller NR, Merritt SA, Klauber-Demore N, Hultman CS, Blau WS. Acute and persistent postoperative pain after breast surgery. Pain Med. 2009 May-Jun;10(4):708-15. doi: 10.1111/j.1526-4637.2009.00611.x. Epub 2009 Apr 22. PMID 19453965
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Stoffels I, Dissemond J, Korber A, Hillen U, Poeppel T, Schadendorf D, Klode J. Reliability and cost-effectiveness of sentinel lymph node excision under local anaesthesia versus general anaesthesia for malignant melanoma: a retrospective analysis in 300 patients with malignant melanoma AJCC Stages I and II. J Eur Acad Dermatol Venereol. 2011 Mar;25(3):306-10. doi: 10.1111/j.1468-3083.2010.03786.x. PMID 20626530
- [Background] Stoffels I, Dissemond J, Schulz A, Hillen U, Schadendorf D, Klode J. Reliability and cost-effectiveness of complete lymph node dissection under tumescent local anaesthesia vs. general anaesthesia: a retrospective analysis in patients with malignant melanoma AJCC stage III. J Eur Acad Dermatol Venereol. 2012 Feb;26(2):200-6. doi: 10.1111/j.1468-3083.2011.04036.x. Epub 2011 Mar 17. PMID 21414036
- [Background] Pawa A, Wight J, Onwochei DN, Vargulescu R, Reed I, Chrisman L, Pushpanathan E, Kothari A, El-Boghdadly K. Combined thoracic paravertebral and pectoral nerve blocks for breast surgery under sedation: a prospective observational case series. Anaesthesia. 2018 Apr;73(4):438-443. doi: 10.1111/anae.14213. Epub 2018 Jan 12. PMID 29327341
- [Background] Woodworth GE, Ivie RMJ, Nelson SM, Walker CM, Maniker RB. Perioperative Breast Analgesia: A Qualitative Review of Anatomy and Regional Techniques. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):609-631. doi: 10.1097/AAP.0000000000000641. PMID 28820803
- [Background] Kwekkeboom K. Postmastectomy pain syndromes. Cancer Nurs. 1996 Feb;19(1):37-43. doi: 10.1097/00002820-199602000-00005. PMID 8904385
- [Background] Vecht CJ, Van de Brand HJ, Wajer OJ. Post-axillary dissection pain in breast cancer due to a lesion of the intercostobrachial nerve. Pain. 1989 Aug;38(2):171-6. doi: 10.1016/0304-3959(89)90235-2. PMID 2780072
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Lee TH, Marcantonio ER, Mangione CM, Thomas EJ, Polanczyk CA, Cook EF, Sugarbaker DJ, Donaldson MC, Poss R, Ho KK, Ludwig LE, Pedan A, Goldman L. Derivation and prospective validation of a simple index for prediction of cardiac risk of major noncardiac surgery. Circulation. 1999 Sep 7;100(10):1043-9. doi: 10.1161/01.cir.100.10.1043. PMID 10477528
- [Background] Jette M, Sidney K, Blumchen G. Metabolic equivalents (METS) in exercise testing, exercise prescription, and evaluation of functional capacity. Clin Cardiol. 1990 Aug;13(8):555-65. doi: 10.1002/clc.4960130809. PMID 2204507
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Franceschini J, Jardim JR, Fernandes AL, Jamnik S, Santoro IL. Reproducibility of the Brazilian Portuguese version of the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire used in conjunction with its lung cancer-specific module. J Bras Pneumol. 2010 Sep-Oct;36(5):595-602. doi: 10.1590/s1806-37132010000500011. English, Portuguese. PMID 21085825
- [Background] Agha RA, Fowler AJ, Rajmohan S, Barai I, Orgill DP; PROCESS Group. Preferred reporting of case series in surgery; the PROCESS guidelines. Int J Surg. 2016 Dec;36(Pt A):319-323. doi: 10.1016/j.ijsu.2016.10.025. Epub 2016 Oct 19. PMID 27770639
- See also: EORTC QLQ-C30 Scoring Manual. 2001 EORTC, Brussels. ISBN 2-9300 64-22-6. — https://www.eortc.org/app/uploads/sites/2/2018/02/SCmanual.pdf